CLINICAL TRIAL: NCT06145308
Title: Cancer Hospital, Chinese Academy of Medical Sciences/National Cancer Center of China
Brief Title: Precision Treatment of Recurrent/Metastatic Salivary Gland Carcinoma Guided by Molecular Typing
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Collaborators: Peking University Hospital of Stomatology (Other)
Responsible Party: Principal Investigator, Fei Ma, Chief physician and deputy chief of internal medicine, Peking Union Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCC4132
Record Dates: First submitted 2023-09-07; First posted 2023-11-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-12

CONDITIONS: Salivary Gland Carcinoma; Precision Therapy
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — Leuprolide; bicalutamide; abiraterone; Platinum; Albumin-Bound Paclitaxel; Carboplatin; apatinib; camrelizumab; Trastuzumab; pyrotinib; darolutamide; Goserelin; pertuzumab; Docetaxel; Fulvestrant; Poly(ADP-ribose) Polymerase Inhibitors; enfortumab vedotin

STUDY DESIGN:
Intervention Model Description: The study employs a master-protocol platform design with the primary objective of identifying promising subgroups; new drug regimens may be added during the trial, while ineffective arms are closed based on interim monitoring. The trial consists of two stages. In Stage 1, each experimental arm uses a Bayesian Optimal Phase II (BOP2) design to assess whether the regimen shows sufficient efficacy to warrant further investigation. Arms demonstrating promising activity proceed to Stage 2（Simon two-stage design）.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (19):
- Cohort 1 (HER2-positive, RC48-ADC) (Experimental): Disitamab vedotin 2.5 mg/kg will be administered as an intravenous infusion every 2 weeks (Q2W) as monotherapy, or in combination with physician-selected platinum-based chemotherapy (carboplatin 200-250 mg/m² IV Q2W or cisplatin 50 mg/m² IV Q2W).
  Interventions: Drug: Cohort 1 (HER2-positive, RC48-ADC)
- Cohort 2 (NTRK-fusion or NTRK-mutant) (Experimental): larotrectinib 100 mg orally twice daily or entrectinib 600 mg orally once daily;
  Interventions: Drug: Cohort 2 (NTRK-fusion or NTRK-mutant)
- Cohort 3 (AR-positive, leuprolide + bicalutamide + abiraterone) (Experimental): leuprolide 3.75 mg subcutaneously every 4 weeks, bicalutamide 50 mg orally once daily, and abiraterone 1 000 mg orally once daily.
  Interventions: Drug: Cohort 3 (AR-positive, leuprolide + bicalutamide + abiraterone)
- Cohort 4 (TROP2 ADC) (Experimental): ESG401 16 mg/kg IV (days 1, 8, 15, q4w), sacituzumab govitecan 10 mg/kg IV (days 1 & 8, q3w), or sacituzumab tirumotecan 5 mg/kg IV q2w.
  Interventions: Drug: TROP2 ADC
- Cohort 5 (ACC-TKI) (Experimental): apatinib 250 mg qd po or anlotinib 12 mg
  Interventions: Drug: TKI
- Cohort 6 (albumin-bound paclitaxel + platinum) (Experimental): albumin-bound paclitaxel 260 mg/m² IV q3w plus physician-selected cisplatin 75 mg/m² IV q3w or carboplatin 350 mg/m² IV q3w.
  Interventions: Drug: Albumin-paclitaxel + platinum
- Cohort 7 (albumin-bound paclitaxel + carboplatin + apatinib + camrelizumab) (Experimental): albumin-bound paclitaxel 260 mg/m² IV q3w, carboplatin 350 mg/m² IV q3w, camrelizumab 200 mg IV q3w, and apatinib 250 mg qd po.
  Interventions: Drug: Albumin-paclitaxel + carboplatin + apatinib + camrelizumab
- Cohort 8 (HER2-positive, albumin-bound paclitaxel + trastuzumab + pyrotinib) (Experimental): albumin-bound paclitaxel 260 mg/m² + trastuzumab (loading 8 mg/kg → 6 mg/kg IV q3w) + pyrotinib 400 mg PO qd.
  Interventions: Drug: albumin-bound paclitaxel+trastuzumab+pyrotinib
- Cohort 9 (HER2-positive, DS-8201 ± pertuzumab) (Experimental): trastuzumab deruxtecan 5.4 mg/kg IV q3w ± pertuzumab (loading 840 mg → 420 mg IV q3w).
  Interventions: Drug: HER2,trastuzumab deruxtecan± pertuzumab
- Cohort 10 (HER2+/AR+, darolutamide + goserelin + pertuzumab + trastuzumab) (Experimental): darolutamide 600 mg PO bid + goserelin 10.8 mg SC q12w + pertuzumab/trastuzumab loading 15 mL → 10 mL SC q3w.
  Interventions: Drug: AR,darolutamide + goserelin+pertuzumab/trastuzumab
- Cohort 11 (AR-positive, darolutamide + goserelin + docetaxel) (Experimental): darolutamide 600 mg PO bid + goserelin 10.8 mg SC q12w + docetaxel 75 mg/m² IV q3w.
  Interventions: Drug: AR,darolutamide +goserelin +docetaxel
- Cohort 12 (ivonescimab) (Experimental): ivonescimab 20 mg/kg + investigator-choice platinum doublet (albumin-paclitaxel 260 mg/m², liposomal paclitaxel 175 mg/m², docetaxel 75 mg/m², or vinorelbine 25 mg/m² d1,d8) plus cisplatin 75 mg/m² or carboplatin AUC 5-6 IV q3w.
  Interventions: Drug: ivonescimab + investigator-choice platinum doublet+
- Cohort 13 (iparomlimab + tuvonralimab) (Experimental): iparomlimab 5 mg/kg + platinum doublet (as above) ± bevacizumab 5 mg/kg IV q3w.
  Interventions: Drug: iparomlimab + tuvonralimab
- Cohort 14 (cadonilimab) (Experimental): cadonilimab 10 mg/kg + platinum doublet (as above) ± bevacizumab 5 mg/kg IV q3w.
  Interventions: Drug: cadonilimab
- Cohort 15 (HR-positive) (Experimental): CDK4/6 inhibitor (abemaciclib 150 mg PO bid or palbociclib 125 mg PO qd) plus AI (letrozole 2.5 mg, anastrozole 1 mg, or exemestane 20 mg PO qd) or fulvestrant 500 mg IM q4w
  Interventions: Drug: CDK4/6 inhibitor+AI or fulvestrant
- Cohort 16 (PI3K-mutant) (Experimental): alpelisib 300 mg PO qd plus fulvestrant 500 mg IM q4w.
  Interventions: Drug: alpelisib+fulvestrant
- Cohort 17 (homologous-recombination-deficient) (Experimental): PARP inhibitor (olaparib 300 mg PO bid, niraparib 300 mg PO qd, fluzoparib 150 mg PO bid, or pamiparib 60 mg PO bid).
  Interventions: Drug: PARP inhibitor
- Cohort 18 (Nectin-4 ADC) (Experimental): enfortumab vedotin 1.25 mg/kg IV d1,d8,d15 (max 125 mg) ± ICI (pembrolizumab 200 mg, camrelizumab 200 mg, or toripalimab 240 mg IV q3w).
  Interventions: Drug: enfortumab vedotin
- Cohort 19 (HER2-positive, pyrotinib + pertuzumab + trastuzumab) (Experimental): pyrotinib 400 mg PO qd + pertuzumab/trastuzumab loading 15 mL → 10 mL SC q3w.
  Interventions: Drug: HER2, pyrotinib + pertuzumab/trastuzumab

INTERVENTIONS:
Drug: Cohort 1 (HER2-positive, RC48-ADC) — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: HER2,Vedolizumab
  Arms: Cohort 1 (HER2-positive, RC48-ADC)
Drug: Cohort 2 (NTRK-fusion or NTRK-mutant) — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: NTRK-inhibitor
  Arms: Cohort 2 (NTRK-fusion or NTRK-mutant)
Drug: Cohort 3 (AR-positive, leuprolide + bicalutamide + abiraterone) — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: AR,leuprolide + bicalutamide + abiraterone
  Arms: Cohort 3 (AR-positive, leuprolide + bicalutamide + abiraterone)
Drug: TROP2 ADC — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 4 (TROP2 ADC)
  Arms: Cohort 4 (TROP2 ADC)
Drug: TKI — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 5 (ACC-TKI)
  Arms: Cohort 5 (ACC-TKI)
Drug: Albumin-paclitaxel + platinum — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 6 (albumin-bound paclitaxel + platinum)
  Arms: Cohort 6 (albumin-bound paclitaxel + platinum)
Drug: Albumin-paclitaxel + carboplatin + apatinib + camrelizumab — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 7 (albumin-bound paclitaxel + carboplatin + apatinib + camrelizumab)
  Arms: Cohort 7 (albumin-bound paclitaxel + carboplatin + apatinib + camrelizumab)
Drug: albumin-bound paclitaxel+trastuzumab+pyrotinib — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort8 (HER2-positive, albumin-bound paclitaxel + trastuzumab + pyrotinib)
  Arms: Cohort 8 (HER2-positive, albumin-bound paclitaxel + trastuzumab + pyrotinib)
Drug: HER2,trastuzumab deruxtecan± pertuzumab — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort9(HER2-positive, DS-8201 ± pertuzumab)
  Arms: Cohort 9 (HER2-positive, DS-8201 ± pertuzumab)
Drug: AR,darolutamide + goserelin+pertuzumab/trastuzumab — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 10 (HER2+/AR+, darolutamide + goserelin + pertuzumab + trastuzumab)
  Arms: Cohort 10 (HER2+/AR+, darolutamide + goserelin + pertuzumab + trastuzumab)
Drug: AR,darolutamide +goserelin +docetaxel — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 11 (AR-positive, darolutamide + goserelin + docetaxel)
  Arms: Cohort 11 (AR-positive, darolutamide + goserelin + docetaxel)
Drug: ivonescimab + investigator-choice platinum doublet+ — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 12 (ivonescimab)
  Arms: Cohort 12 (ivonescimab)
Drug: iparomlimab + tuvonralimab — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 13 (iparomlimab + tuvonralimab)
  Arms: Cohort 13 (iparomlimab + tuvonralimab)
Drug: cadonilimab — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 14 (cadonilimab)
  Arms: Cohort 14 (cadonilimab)
Drug: CDK4/6 inhibitor+AI or fulvestrant — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 15 (HR-positive)
  Arms: Cohort 15 (HR-positive)
Drug: alpelisib+fulvestrant — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 16 (PI3K-mutant)
  Arms: Cohort 16 (PI3K-mutant)
Drug: PARP inhibitor — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 17 (homologous-recombination-deficient)
  Arms: Cohort 17 (homologous-recombination-deficient)
Drug: enfortumab vedotin — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 18 (Nectin-4 ADC)
  Arms: Cohort 18 (Nectin-4 ADC)
Drug: HER2, pyrotinib + pertuzumab/trastuzumab — Neoadjuvant / conversion phase: After 2-6 cycles of protocol therapy, patients are re-evaluated. Those deemed resectable undergo surgery of the primary tumour ± metastatic sites, followed by radiotherapy or other modalities (e.g., radiofrequency ablation) at the investigator's discretion. Patients who remain unresectable after six cycles continue the same regimen until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to stop.
  Adjuvant phase: Treatment is administered for 2 years, or until intolerable toxicity or withdrawal of consent.
  Salvage phase: Therapy continues until disease progression, intolerable toxicity, withdrawal of consent, or investigator decision to terminate.
  Other Names: Cohort 19 (HER2-positive, pyrotinib + pertuzumab + trastuzumab)
  Arms: Cohort 19 (HER2-positive, pyrotinib + pertuzumab + trastuzumab)

SUMMARY:
Patients with salivary gland carcinoma were divided into groups according to HER2, NTRK, AR, TROP-2, etc. Patients in different groups were given precision targeted therapy or chemotherapy to evaluate the efficacy (ORR rate) and safety of precision therapy.

DETAILED DESCRIPTION:
Patients with locally advanced/recurrent or oligometastatic salivary gland carcinoma will be stratified by HER2, NTRK, AR, TROP-2, etc., and receive precision-targeted or chemotherapy regimens, with efficacy (objective response rate, etc.) and safety of neoadjuvant/conversion therapy evaluated.

To assess the efficacy of post-operative adjuvant therapy guided by minimal residual disease (MRD) testing in locally advanced salivary gland carcinoma.

Patients with locally advanced/recurrent or symptomatic, rapidly progressive metastatic salivary gland carcinoma who are intolerant of or refuse surgery and radiotherapy will be molecularly stratified and treated with precision regimens, with efficacy (objective response rate, etc.) and safety of salvage therapy evaluated.

To evaluate efficacy (objective response rate, etc.) and safety of later-line therapy for locally advanced/recurrent or distant metastatic salivary gland carcinoma.

Using multi-omic approaches to explore salivary gland carcinoma heterogeneity and biomarkers associated with recurrence, metastasis, treatment response and prognosis.

To investigate concordance between drug-sensitivity testing using ex-vivo 3D tumour models and actual clinical outcomes, and to guide later-line treatment selection based on drug-sensitivity results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologic diagnosis of salivary gland carcinoma

  * The tumor tissues were subjected to HER2/NTRK/AR/TROP-2 immunohistochemical staining.

    * ECOG physical status 0 or 1 score in the 3 days before the first medication of the study treatment;

      * Age 18 or older - no upper limit;

        * Life expectancy is more than 3 months; ⑥Have at least one measurable lesion according to RECIST1.1 standards; ⑦Women of childbearing age must have a negative pregnancy test within 7 days before the first medication, and agree to receive the necessary contraceptive measures;

          ⑧The patient must have adequate liver, kidney, bone marrow, heart and lung and other organ functions:

          ⑨Understanding and voluntarily signing informed consent prior to performing any research-related evaluation/operation;

          ⑩Ability to comply with research visit schedules and other programmatic requirements.

Exclusion Criteria:

* Known hypersensitivity or delayed anaphylaxis to any agents in this trial;

  * Major surgery had been performed within 4 weeks prior to the start of the study and did not fully recover;

    * Have received a live vaccine within 4 weeks before the start of the study or plan to receive any vaccine during the study period ;

      * To study the occurrence of arterial/venous thrombosis events within 6 months before medication;

        * Major cardiovascular diseases;

          * Is suffering from uncontrolled systemic diseases, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, cirrhosis, etc.;

            * Is suffering from an active infection that requires systemic treatment;

              * History of active tuberculosis; ⑨ Positive human immunodeficiency virus (HIV) test result; ⑩ Patients with chronic hepatitis B or active hepatitis C. ⑪Conditions that the investigator believes will affect the safety or compliance of the drug therapy in this study ⑫Female/male who is pregnant or breastfeeding or who intends to give birth;

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2028-07-10 (Estimated)

PRIMARY OUTCOMES:
ORR | ORR at the end of Cycle 2 (each cycle is 21 days)
  ORR rates for neoadjuvant and translational therapy in patients with locally advanced/recurrent and advanced oligometastatic salivary gland cancer and ORR rate of salvage therapy for locally advanced/recurrent or distantly metastatic salivary gland carcinoma with rapid progression that cannot tolerate or refuses surgery

SECONDARY OUTCOMES:
MPR; | MPR rate at the end of surgical treatment
  MPR rates in patients who received neoadjuvant and translational therapy and then underwent surgery
R0 resection rate; | R0 resection rate at the end of surgical treatment
  R0 resection rate in patients who received neoadjuvant and translational therapy and then underwent surgery
Facial nerve protection rate | Facial nerve protection rate at the end of surgical treatment
  Facial nerve protection rate in patients who received neoadjuvant and translational therapy and then underwent surgery
DFS | DFS rates at 3-year
  3-year DFS rates for patients who underwent surgery
PFS; | PFS Rate at 2-Year
  2-Year PFS Rate for Patients Receiving Rescue Therapy
OS | OS rate at 5-year
  OS for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhang, Principal Investigator — Department of Oral and Maxillofacial Surgery, Peking University School and Hospital of Stomatology
Locations (2):
- China (2):
  - Fei Ma, Beijing, Beijing Municipality
  - National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing

IPD SHARING:
Plan to Share IPD: No